CLINICAL TRIAL: NCT03584711
Title: A Phase II Study Evaluating FOLFOX + Panitumumab According to a "Stop and go" Strategy With a Reintroduction Loop After Progression on Fluoropyrimidine as Maintenance Treatment, as the First Line in Patients With Metastatic Colorectal Adenocarcinoma Without a RAS Mutation
Brief Title: FOLFOX + Panitumumab According to a "Stop and go" Strategy With a Reintroduction Loop After Progression on Fluoropyrimidine as Maintenance Treatment, as the First Line in Patients With Metastatic Colorectal Adenocarcinoma Without a RAS Mutation
Acronym: OPTIPRIME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FFCD 1605
Record Dates: First submitted 2018-06-19; First posted 2018-07-12 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Stop and Go strategy; RAS Wild-type
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Folfox protocol; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FOLFOX + panitumumab (Experimental): 1 cylce every 14 days : Panitumumab : 6 mg/kg en IV (J1) during 60 minutes for 1st infusion followed by 30 to 60 minutes Oxaliplatine : 85 mg/m² inG5% orNaCl 0.9% in IV (D1) during 2 hours Acide folinique : 400 mg/m² (or200 mg/m² if Elvorine) in IV (D1) 5Fu bolus : 400 mg/m² in IV 5FU continu : 2400 mg/m² in IV during 46 hours
  LV5FU2 : 1 cycle every 14 days Acide folinique : 400 mg/m² (or 200 mg/m² ifElvorine) in IV (D1) during 2 hours 5FU bolus : 400 mg/m² in IV 5FU continu : 2400 mg/m² in IV during 46 hours
  Interventions: Combination Product: FOLFOX + panitumumab

INTERVENTIONS:
Combination Product: FOLFOX + panitumumab — FOLFOX + panitumumab according to a "stop and go" strategy with a reintroduction loop after progression on fluoropyrimidine as maintenance treatment

SUMMARY:
Single-arm, multi-centre phase II study The primary objective is to evaluate the time to failure of the strategy.

DETAILED DESCRIPTION:
The purpose of the OPTIPRIME phase II non-randomised study is to evaluate the efficacy and tolerability of the combination of FOLFOX plus panitumumab according to a "stop and go" strategy. If disease control is achieved while on induction treatment, oxaliplatin and panitumumab will be stopped after the sixth cycle; a maintenance treatment of fluoropyrimidine alone will be continued. In case of progression during maintenance treatment, oxaliplatin and panitumumab reintroduction loops will take place according to the same regimen (maintenance treatment after six cycles of the reintroduced therapy if disease control is achieved).

ELIGIBILITY:
Inclusion Criteria:

* - Histologically proven colorectal adenocarcinoma without RAS mutation
* Confirmed, non-resectable metastatic disease (Stage IV)
* No prior chemotherapy except perioperative or adjuvant chemotherapy discontinued for more than 12 months
* At least one measurable metastasis according to the RECIST v1.1 criteria
* Age ≥ 18 years
* WHO ≤ 2
* Neutrophils > 1500 /mm3, platelets> 100 000/mm3, Hb > 9 g/dL
* Creatinine clearance > 50 mL/min according to the MDRD formula
* Serum bilirubin < 25 µmol/L, AST, ALT, Alk Phos < 2.5 x ULN or < 5 x ULN in case of liver metastases
* PT > 60%, albumin ≥ 25g/L
* Estimated life expectancy ≥ 3 months
* Patient affiliated to a social security scheme
* Patient informed and informed consent form signed

Exclusion Criteria:

* - Presence of uncontrolled symptomatic brain metastases
* RAS mutation (KRAS or NRAS mutation)
* Patient taking warfarin. If treated with anticoagulant at the indicated effective dose, this must be replaced with low molecular weight heparin before inclusion
* Known DPD deficiency
* Peripheral neuropathy > 1 (NCI CTCAE v4.0)
* Patient with interstitial pneumonitis or pulmonary fibrosis
* History of chronic diarrhoea or inflammatory disease of the colon or rectum, or obstruction or sub-obstruction during symptomatic treatment
* Poorly controlled chronic skin disease
* Any known specific contraindication or allergy to the medicinal products used in the study
* Patient simultaneously included in another clinical trial involving an investigational drug (example: chemotherapy, targeted therapy, immunotherapy)
* Arterial hypertension not controlled by medical treatment (Systolic BP ≥ 160 mmHg end/or diastolic BP ≥ 90 mmHg)
* Any progressive pathology not stabilised over the past 6 months: hepatic failure, renal failure, respiratory failure
* The following conditions in the 6 months prior to inclusion: myocardial infarction, severe/unstable angina, coronary artery bypass surgery, congestive heart failure NYHA class II, III or IV, stroke or transient ischaemic attack
* Patient who has received a transplant, is seropositive for HIV, hepatitis B or hepatitis C or has other immunodeficiency syndromes
* History of malignant pathologies during the past 5 years except basal cell carcinoma of the skin or cervical carcinoma in situ, properly treated
* QT/QTc interval > 450 msec for men and > 470 msec for women
* K+ < LNL, Mg2+ < LNL, Ca2+ < LNL
* Lack of effective contraception in patients (men and/or women) of childbearing age, pregnant or breastfeeding women, women of childbearing age who have not had a pregnancy test
* Persons in custody or under wardship
* Impossibility of undergoing medical monitoring during the trial for geographical, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Time to failure of the strategy | Up to 20 months
  Time to strategy Failure is defined as the time from date of inclusion to strategy failure (Radiological progression under treatment or death or definitive treatment discontinuation or recurrence after curative surgery with or without adjuvant treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste Bachet, Pr, Principal Investigator — Federation Francophone de Cancerologie Digestive
Locations (118):
- France (117):
  - Clinique Trenel, Sainte-Colombe, Lyon
  - Clinique Claude Bernard, Albi
  - Hopital Sud, Amiens
  - Clinique de L'Europe, Amiens
  - CHU Amiens Picardie Hôpital Sud, Amiens
  - Clinique de l'Europe, Amiens
  - Chu D'Angers, Angers
  - CHU, Angers
  - Hopital Prive D'Antony, Antony
  - Hôpital Privé, Antony
  - Centre Marie Curie, Arras
  - Hopital Les Bonnettes, Arras
  - Hôpital Privé Les Bonnettes, Arras
  - CH Henri Duffaut, Avignon
  - Institut Sainte Catherine, Avignon
  - Ch Cote Basque, Bayonne
  - Centre Hospitalier Côte Basque, Bayonne
  - Ch de Beauvais, Beauvais
  - Centre Hospitalier, Beauvais
  - Ch de Beziers Cedex, Béziers
  - Centre Hospitalier, Béziers
  - Polyclinique Saint Privat, Boujan-sur-Libron
  - Cmco Cote D'Opale, Boulogne-sur-Mer
  - Hopital Duchenne, Boulogne-sur-Mer
  - Hôpital Duchenne, Boulogne-sur-Mer
  - Hopital Morvan - Chu, Brest
  - CHU, Brest
  - Centre Francois Baclesse, Caen
  - Centre François Baclesse, Caen
  - Ch Cahors, Cahors
  - Loire Vendee Ocean, Challans
  - Hôpital Louis Pasteur, Chartres
  - Centre Hospitalier General, Châlons-en-Champagne
  - Centre Hospitalier, Châlons-en-Champagne
  - Ch de Cholet, Cholet
  - Centre Hospitalier, Cholet
  - Hopitaux Civils de Colmar, Colmar
  - Hôpitaux Civils de Colmar, Colmar
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Clinique de Flandre, Coudekerque-Branche
  - Service de Medecine, Digne-les-Bains
  - Centre Hospitalier, Digne-les-Bains
  - Centre G. François Leclerc, Dijon
  - CHU, Dijon
  - CH, Dunkirk
  - Centre Hospitalier, Dunkirk
  - Hopital Jacques Monod, Flers
  - CH J Monod, Flers
  - CHU Martanique Hôpital Clarac, FORT de France
  - Chi de Frejus Saint-Raphael, Fréjus
  - CHI Fréjus St Raphaël, Fréjus
  - Hôpital Michallon, Grenoble
  - Polyclinique de Blois - 3Eme Etage, La Chaussée-Saint-Victor
  - Polyclinique Blois, La Chaussée-Saint-Victor
  - Chd Vendee, La Roche-sur-Yon
  - CHD VENDEE (Les Oudairies), La Roche-sur-Yon
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Ch Du Mans, Le Mans
  - Centre Hospitalier, Le Mans
  - Centre Hospitalier Schaffner, Lens
  - Centre Hospitalier, Lens
  - Chru Hopital Claude Huriez 4Eme Est, Lille
  - CHU Claude Huriez, Lille
  - Hôpital Privé LE BOIS, Lille
  - Ch St Joseph-St Luc, Lyon
  - CH Saint Joseph St Luc, Lyon
  - Prive - Jean Mermoz, Lyon
  - Chi F. Quesnay, Mantes-la-Jolie
  - Hopital Europeen Marseille, Marseille
  - Hôpital Européen, Marseille
  - Ch de Meaux, Meaux
  - Centre Hospitalier, Meaux
  - Hopital Layne, Mont-de-Marsan
  - Centre Hospitalier, Montélimar
  - CHI, Montfermeil
  - Polyclinique de Gentilly, Nancy
  - Centre d'oncologie de Gentilly, Nancy
  - Hopital Prive Du Confluent Sas, Nantes
  - Le Confluent SAS, Nantes
  - Ch de Niort - Sce D'Oncologie, Niort
  - Centre Hospitalier, Niort
  - CHR, Orléans
  - Chu Cochin, Paris
  - Groupe Hospitalier Pitie-Salpetriere, Paris
  - CHU Bichat, Paris
  - Groupe Diaconnesses Croix St Simon, Paris
  - HEGP, Paris
  - Hôpital Cochin (APHP), Paris
  - La Pitie Salpetriere, Paris
  - Hôpital Haut Lévêque, Pessac
  - Centre Hospitalier, Périgueux
  - Polyclinique Francheville, Périgueux
  - CHU, Poitiers
  - Clinique de la Croix du Sud, Quint-Fonsegrives
  - Polyclinique de Courlancy, Reims
  - Institut du Cancer Courlancy, Reims
  - CH de Romans, Romans-sur-Isère
  - Centre Hospitalier, Roubaix
  - CHU, Rouen
  - Saint Hilaire - Privee, Rouen
  - CHP, Saint-Grégoire
  - Clinique de l'Union, Saint-Jean
  - Centre Médical Côte d'Opale, Saint-Martin-Boulogne
  - Hopital Nord Chu Saint Etienne, Saint-Priest-en-Jarez
  - Centre Hospitalier, Saint-Quentin
  - Clinique Trenel, Sainte-Colombe
  - Clinique Charcot, Sainte-Foy-lès-Lyon
  - Clinique Ste Anne, Strasbourg
  - Centre Paul Strauss, Strasbourg
  - Clinique Sainte Anne, Strasbourg
  - Polyclinique de L'Ormeau, Tarbes
  - Hôpital Sainte Musse, Toulon
  - Clinique Pasteur, Toulouse
  - CHRU, Tours
  - Clinique des Dentellières, Valenciennes
  - Hôpital Privé, Villeneuve-d'Ascq
  - Médipôle Hôpital Mutualiste Lyon Villeurbanne, Villeurbanne
- Chu de Fort de France, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: Undecided